CLINICAL TRIAL: NCT05833347
Title: Evaluation of Difficult Laryngoscopy With Ultrasonography in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Osman Kaya, Trainee, Eskisehir Osmangazi University
Other Study IDs: ESOGU-OKAYA-001
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-11

CONDITIONS: Intubation; Difficult or Failed; Difficult Laryngoscopy
Keywords: Difficult laryngoscopy; Ultrasonography; Pediatric Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2-8 Years Paediatric Patients: During the preoperative evaluation, demographic data and airway physical examination results (Mallampati score) of the patients will be recorded. Patients who have received preoperative sedation will be positioned supine on the operating table, and ultrasound-guided measurements of soft tissue distances will be taken using a linear probe with a frequency range of 6-13 Hz. The distance between the hyoid bone and skin (DSHB), distance between the vocal cord anterior commissure and skin (DSAC), and distance between the epiglottis and skin (DSE) will be measured. The A/E (Anterior Commissura/Epiglottis) ratio will be calculated after measurements.
  After standard monitoring and anesthesia induction, difficult laryngoscopy will be evaluated using the Modified Cormack Lehane Score, which grades the visibility of vocal cords and glottic structures. A grade of 3 or 4 on this scale will be considered as difficult laryngoscopy and recorded as such.
  Interventions: Diagnostic Test: Distance between Skin-Hyoid Bone(DSHB); Diagnostic Test: Distance between Skin-Vocal Cord Anterior Commissura(DSAC); Diagnostic Test: Distance between Skin-Epiglottic(DSE)

INTERVENTIONS:
Diagnostic Test: Distance between Skin-Hyoid Bone(DSHB) — Hyoid bone-skin distance Other Name: DSHB
Diagnostic Test: Distance between Skin-Vocal Cord Anterior Commissura(DSAC) — Vocal cord anterior commissura-skin distance Other Name: DSAC
Diagnostic Test: Distance between Skin-Epiglottic(DSE) — Skin-epiglottic distance Other Name: DSE

SUMMARY:
Pediatric patients pose challenges in airway management due to anatomical and physiological changes. Using recommended predictive tests for predicting difficult airway can be improved by combining them with ultrasound measurement of the anterior soft tissues of the neck. In this study, the investigators aim to evaluate the ultrasound measurement of anterior neck soft tissues in paediatric patients before anesthesia induction, to anticipate difficult laryngoscopy.

DETAILED DESCRIPTION:
Eligible participants for this study will be patients aged 2-8 years scheduled for elective surgery under general anesthesia who have provided informed consent. During the preoperative evaluation, demographic data and airway physical examination results (Mallampati score) of the patients will be recorded. Patients who have received preoperative sedation will be positioned supine on the operating table, and ultrasound-guided measurements of soft tissue distances will be taken using a linear probe with a frequency range of 6-13 Hz. The distance between the hyoid bone and skin (DSHB), distance between the vocal cord anterior commissure and skin (DSAC), and distance between the epiglottis and skin (DSE) will be measured. The A/E (Anterior Commissura/Epiglottis) ratio will be calculated after measurements.

After standard monitoring and anesthesia induction, difficult laryngoscopy will be evaluated using the Modified Cormack Lehane Score, which grades the visibility of vocal cords and glottic structures. A grade of 3 or 4 on this scale will be considered as difficult laryngoscopy and recorded as such. Tracheal intubation will be performed by an anesthesiologist with at least two years of experience who is unaware of the ultrasound measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo general anesthesia for elective surgery
* American Anesthesiology Association physical classification (ASA) status I-III
* Body mass index (BMI) above 30

Exclusion Criteria:

* Patients with a history of difficult airway or with conditions that are known to be associated with a difficult airway, such as syndromic or metabolic diseases.
* Patients with congenital maxillofacial defects.
* Patients with tracheal or laryngeal pathology.
* Patients with pulmonary diseases such as bronchial asthma or airway hyperreactivity.
* Patients with allergies to ultrasound gel.
* Patients with weight percentile outside the range of 10-90 percentiles.
* Patients undergoing emergency surgery.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A hundred twenty patients, aged 2-8 years-old, with an American Anesthesiology Association physical classification (ASA) I-III planned to undergo general anesthesia for elective surgery, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy | 1 minute
  As the primary outcome, correlation of distance between the hyoid bone and skin (DSHB), distance between the vocal cord anterior commissure and skin (DSAC), and distance between the epiglottis and skin (DSE) and A/E (Anterior Commissura/Epiglottis) ratio with the Cormack Lehane score will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Kaya, Res Assist., Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Wu J, Dong J, Ding Y, Zheng J. Role of anterior neck soft tissue quantifications by ultrasound in predicting difficult laryngoscopy. Med Sci Monit. 2014 Nov 18;20:2343-50. doi: 10.12659/MSM.891037. PMID 25403231
- [Background] Alessandri F, Antenucci G, Piervincenzi E, Buonopane C, Bellucci R, Andreoli C, Alunni Fegatelli D, Ranieri MV, Bilotta F. Ultrasound as a new tool in the assessment of airway difficulties: An observational study. Eur J Anaesthesiol. 2019 Jul;36(7):509-515. doi: 10.1097/EJA.0000000000000989. PMID 31742568
- [Background] Altun D, Kara H, Bozbora E, Ali A, Dinc T, Sonmez S, Buget M, Aydemir L, Basaran B, Tugrul M, Camci E. The Role of Indirect Laryngoscopy, Clinical and Ultrasonographic Assessment in Prediction of Difficult Airway. Laryngoscope. 2021 Feb;131(2):E555-E560. doi: 10.1002/lary.28849. Epub 2020 Jul 30. PMID 32730647